CLINICAL TRIAL: NCT04967495
Title: Transarterial Chemoembolization Combined With Lenvatinib and Iodion-125 Seeds Brachytherapy for Hepatocellular Carcinoma With Portal Vein Branch Tumor Thrombus: a Single Center, Prospective, Randomized Control Trail
Brief Title: TACE Plus Multikinase Inhibitor and I-125 Seeds Brachytherapy for HCC With Branch PVTT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-07
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular Carcinoma; Transarterial chemoembolization; Tyrosine kinase inhibitor; iodion-125 seed
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE-Len-I (Experimental): TACE combined with lenvatinib and iodion-125 seeds brachytherapy
  Interventions: Procedure: TACE combined with lenvatinib and iodion-125 seeds brachytherapy
- TACE-Len (Active Comparator): TACE combined with lenvatinib
  Interventions: Procedure: TACE combined with lenvatinib

INTERVENTIONS:
Procedure: TACE combined with lenvatinib and iodion-125 seeds brachytherapy — TACE will be performed for the patients after randomization. Lenvatinib (body weight ≥ 60 kg, 12mg P.O. QD; body weight < 60 kg, 8mg P.O. QD) will be started at 3-7 days after the first TACE and last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. Iodion-125 seeds will be implanted into the PVTT under CT guidance within 14 days after the first TACE. TACE and iodion-125 seeds implantation can be repeated on demand during follow-up based on the evaluation of laboratory and imaging examination.
  Arms: TACE-Len-I
Procedure: TACE combined with lenvatinib — TACE will be performed for the patients after randomization and it can be repeated on demand during follow-up based on the evaluation of laboratory and imaging examination. Lenvatinib (body weight ≥ 60 kg, 12mg P.O. QD; body weight < 60 kg, 8mg P.O. QD) will be started at 3-7 days after the first TACE and last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first.
  Arms: TACE-Len

SUMMARY:
This study is conducted to evaluate the efficacy and safety of transarterial chemoembolization (TACE) combined with lenvatinib and iodion-125 seeds brachytherapy (TACE-Len-I) compared with TACE combined with lenvatinib (TACE-Len) for hepatocellular carcinoma (HCC) with portal vein branch tumor thrombus (branch PVTT).

DETAILED DESCRIPTION:
This is an single center, randomized controlled trial to evaluate the efficacy and safety of TACE-Len-I compared with TACE-Len for the treatment of HCC with branch PVTT.

171 HCC patients with branch PVTT will be enrolled in this study. The Patients will be treated with TACE-Len-I or TACE-Len using an 2:1 randomization scheme.

TACE will be performed for the patients after randomization. Lenvatinib (body weight ≥ 60 kg, 12mg P.O. QD; body weight < 60 kg, 8mg P.O. QD) will be started at 3-7 days after the first TACE and last until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first. For patients in the TACE-Len-I arm, iodion-125 seeds will be implanted into the PVTT (according to the pre-operative planning) under CT guidance within 14 days after the first TACE. TACE and iodion-125 seeds implantation can be repeated on demand during follow-up based on the evaluation of laboratory and imaging examination.

ELIGIBILITY:
Inclusion Criteria:

1. Age between18 and 75 years.
2. HCC confirmed by histopathology and/or cytology, or diagnosed clinically.
3. Accompanied with tumor thrombus involving unilateral portal vein branch.
4. Child-Pugh class A or B.
5. Eastern Cooperative Group performance status (ECOG) score of 0-2.
6. Serum bilirubin ≤ 51.3 μmol/L, albumin ≥ 28g/L, ALT and AST ≤ 5 times of the upper normal limit, and creatinine ≤ 20g/L.
7. Prothrombin time prolonged for less than 4s or international normalized ratio < 1.7.
8. Neutrophilic granulocyte count ≥ 1.5×10^9/L, platelet count ≥ 50×10^9/L, and hemoglobin level ≥ 85g/L;
9. At least one measurable intrahepatic target lesion.
10. Life expectancy of at least 3 months.

Exclusion Criteria:

1. Diffuse HCC.
2. Extrahepatic metastasis.
3. Tumor thrombus involving both the left and right branch of portal vein or main portal vein.
4. Hepatic vein and/or vena cava invasion.
5. History of organ or cells transplantation.
6. Previous treatment with TACE, intra-arterial infusion chemotherapy, radiotherapy or systemic therapy.
7. History of other malignancies.
8. Serious medical comorbidities.
9. Female patients who are pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2025-01-08 (Estimated); Study Completion 2025-01-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years.
  The time from date of randomization to death due to any cause.

SECONDARY OUTCOMES:
Adverse events (AEs) | 2 years.
  Number of patients with AE, treatment-related AE (TRAE), AE of special interest (AESI), serious adverse event (SAE), assessed by NCI CTCAE v5.0.
Progression free survival (PFS) assessed by investigators according to Modified Response Evalutaion Criteria in Solid Tumors (mRECIST) | 2 years.
  The time from date of randomization until the first occurrence of disease progression (PD) or death due to any cause, whichever occurs first.
Objective response rate (ORR) assessed by investigators according to mRECIST | 2 years.
  The percentage of patients who had a best overall tumor response rating of complete response (CR) or partial response (PR).
Disease control rate (DCR) assessed by investigators according to mRECIST | 2 years.
  The percentage of patients who had a tumor response rating of CR, PR, or stable disease (SD).
Duration of portal patency | 2 years.
  The time from randomization until the date that complete portal vein occlusion was confirmed.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China